CLINICAL TRIAL: NCT05670015
Title: Ocular Changes After Selective Alpha-2 Receptor Agonist.
Brief Title: Ocular Changes With Alpha-2 Receptor Agonist.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Assistant professor of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-2-2023
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma, Suspect; Aberration, Corneal Wavefront
Keywords: Glaucoma suspect; Post-lasik
MeSH Terms: conditions — Ocular Hypertension; Corneal Wavefront Aberration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glaucoma suspect group (Active Comparator): Cases diagnosed as glaucoma suspect
  Interventions: Drug: Low dosage selective alpha-2 receptor agonists topical eyedrop; Drug: High dosage selective alpha-2 receptor agonists topical eyedrop
- Post-refractive surgery group (Active Comparator): Cases had undergone refractive surgery
  Interventions: Drug: Low dosage selective alpha-2 receptor agonists topical eyedrop; Drug: High dosage selective alpha-2 receptor agonists topical eyedrop

INTERVENTIONS:
Drug: Low dosage selective alpha-2 receptor agonists topical eyedrop — Using selective alpha-2 receptor agonists eyedrop in both groups with 0.2% concentration.
  Other Names: Topical selective alpha-2 receptor agonists
Drug: High dosage selective alpha-2 receptor agonists topical eyedrop — Using selective alpha-2 receptor agonists eyedrop in both groups with 0.02% concentration.
  Other Names: Topical selective alpha-2 receptor agonists

SUMMARY:
selective alpha-2 receptor agonists cause changes in intraocular pressure and pupillary size thus may affect patient quality of life.

DETAILED DESCRIPTION:
In this research, we will analyze the effect of selective alpha-2 receptor agonists on the human eye and investigate ocular changes over 6 months after its topical use.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma suspect cases.
* post-refractive surgery cases.

Exclusion Criteria:

* Cases with prostatic hyperplasia or diabetics that may alter the measurements of pupillary diameter.
* Cases with previous history of any retinal intervention or other drugs that may alter intraocular pressure measurements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-10 (Estimated); Study Completion 2023-09-22 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Baseline and 6 months after regular use of the topical eyedrops
  Changes in intraocular pressure measured in mmHg by applanation tonometry

SECONDARY OUTCOMES:
Pupillary diameter | Baseline and 6 months after regular use of the topical eyedrops
  Changes in the pupillary diameter measured in mm by handheld pupillometer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: No